CLINICAL TRIAL: NCT05910060
Title: Ankle Trauma in Children, Application of Ottawa Ankle Rules From 5 Years Old, What is the Impact
Acronym: OTTAWAKIDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GATIN Amélie, Pediatrician, Central Hospital, Nancy, France
Other Study IDs: 2022PI174
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Sports Injuries in Children
Keywords: ankle children Ottawa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- before protocol: patients between 5 and 18 years of age consulting the paediatric emergency department for ankle trauma, before protocol implementation.
- after protocol: patients between 5 and 18 years of age consulting the paediatric emergency department for ankle trauma, after the implementation of the protocol
  Interventions: Diagnostic Test: OTTAWA ANKLE RULES

INTERVENTIONS:
Diagnostic Test: OTTAWA ANKLE RULES — count the ottawa score and do an x-ray if the score is greater than or equal to 1
  Groups: after protocol

SUMMARY:
Ankle sprain in children is a very common pathology. Currently in France, a standard X-ray is done in almost all cases. However, the literature has for several years validated the consideration of the Ottawa ankle rules in children to avoid the realization of these X-rays.

Our study is an evaluation of clinical practice. The aim is to assess the impact of the implementation of a new protocol using the Ottawa ankle rules from the age of 5. In particular, radiographic sparing and absence of diagnostic error.

DETAILED DESCRIPTION:
Main objective: To compare the rate of X-rays performed before and after implementation of the protocol in pediatric emergencies.

Secondary objectives (if applicable):

* Compare the time spent in the emergency room of patients before and after implementation of the protocol
* Evaluate the gain in terms of cost for the healthcare system
* Evaluate the adherence of caregivers to compliance with the protocol
* Evaluate the decrease in the rate of X-rays performed in different age groups.
* Evaluation of the consultation rate in the month for the same reason

Primary endpoint = X-ray rate as a % of X-rays performed on the number of children presenting to pediatric emergencies over the period studied (before implementation of the protocol in a similar period = May to October 2022 / after implementation of the protocol = May to October 2023) Secondary endpoints =

* Time spent in the emergency room in min
* Estimation of the cost for the healthcare system by taking the cost of an x-ray and evaluating the gain on the reduction in the rate of x-rays performed (number of x-rays - cost of an x-ray)
* Evaluation of caregiver compliance by measuring the number of X-rays performed outside the protocol (X-ray performed despite the absence of Ottawa criteria)
* X-ray rate by age group
* Spontaneous reconsultation rate within 1 month

ELIGIBILITY:
Inclusion Criteria:

* 5 to 18 years old
* consulting in pediatric emergency in Nancy children hospital
* for ankle injury

Exclusion Criteria:

Constitutional bone disease Polytrauma Inability to assess the patient (inebriated, altered consciousness, neurosensitive disease, intoxication) Non-acquired walking Injury more than 10 days old Patient re-consults for the same injury previously assessed in the same centre Patient with previous radiographs prior to consultation Open fracture Sensory or vascular deficit Haemophilia Metabolic disease with proven osteopenia

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 5 to 18 years old consulting in pediatric emergency in Nancy children hospital for ankle injury
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
COMPARISON of the rate of x-rays | 4 month
  COMPARISON of the rate of x-rays as a % of x-rays performed among the number of children presenting to paediatric emergency departments over the period studied before and after implementation of the protoc

CONTACTS AND LOCATIONS:
Overall Officials: Amélie GATIN, MD, Principal Investigator — Central Hospital, Nancy, France; Ethan JEOL, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- children hospital Nancy, Vandœuvre-lès-Nancy, Meurthe-et-Moselle, France

IPD SHARING:
Plan to Share IPD: No